CLINICAL TRIAL: NCT00260962
Title: Olanzapine in the Treatment of Low Weight and Obsessional Thinking Among Those With Anorexia Nervosa: A Double Blind Placebo Controlled Study
Brief Title: Olanzapine in the Treatment of Patients With Anorexia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000210-01H; F1D-CA-O092 (Other: Eli Lilly)
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Anorexia Nervosa
Keywords: Pilot Project,; Clinical Trial,; Treatment Outcome,; Psychopharmacology
MeSH Terms: conditions — Anorexia Nervosa | interventions — Olanzapine; Patient Readmission

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo and Treatment as usual (Day Hospital Program). After a 2-week baseline period, placebo was administered for 10 weeks (weeks 3-12 of the study). Day hospital program involved attendance 4 days a week from 9:00 am to 6:00 pm for 12 to 14 weeks, and supervised meals and group therapy.
  Interventions: Behavioral: Day Hospital
- Olanzapine Plus Day Hospital (Experimental): After a 2-week baseline period, Olanzapine was administered for 10 weeks (weeks 3-12 of the study). Olanzapine was prescribed according to a flexible dose regimen, starting at the minimum dose of 2.5 mg/day and titrated slowly by increments of 2.5 mg/week to a maximum dose of 10 mg/day. Day hospital program involved attendance 4 days a week from 9:00 am to 6:00 pm for 12 to 14 weeks, and supervised meals and group therapy.
  Interventions: Drug: Olanzapine; Behavioral: Day Hospital

INTERVENTIONS:
Drug: Olanzapine — After a 2-week baseline period, olanzapine was administered for 10 weeks (weeks 3-12 of the study). Olanzapine was prescribed according to a flexible dose regimen, starting at the minimum dose of at 2.5 mg/day and titrated slowly by increments of 2.5 mg/week to a maximum dose of of 10 mg/day.
  Other Names: Zyprexa
  Arms: Olanzapine Plus Day Hospital
Behavioral: Day Hospital — Day hospital program involved attendance 4 days a week from 9:00 am to 6:00 pm for 12 to 14 weeks, and supervised meals and group therapy.

SUMMARY:
The purpose of the study is to evaluate the efficacy of an anti-psychotic medication, Olanzapine, in achieving desired weight gain in patients identified as having Anorexia Nervosa, either restricting or binge/purge subtype. The study will also evaluate the possible beneficial effects of Olanzapine in reducing the severity of the obsessive and/or anxiety symptoms associated with this disorder.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy of an anti-psychotic medication, Olanzapine, in achieving desired weight gain in patients identified as having Anorexia Nervosa, either restricting or binge/purge subtype. The study will also evaluate the possible beneficial effects of Olanzapine in reducing the severity of the obsessive and/or anxiety symptoms associated with this disorder.

ELIGIBILITY:
Inclusion Criteria:

* those who meet DSM IV criteria of Anorexia Nervosa- either restricting or binge/purge subtype

Exclusion Criteria:

* patients who are actively self destructive and/or suicidal
* patients whose medical status is seriously compromised
* patients whose eating disorder is superimposed on a major psychiatric disorder such as schizophrenia, major affective disorders, dissociative disorder or an active substance abuse disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-09; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H Bissada, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bissada H, Tasca GA, Barber AM, Bradwejn J. Olanzapine in the treatment of low body weight and obsessive thinking in women with anorexia nervosa: a randomized, double-blind, placebo-controlled trial. Am J Psychiatry. 2008 Oct;165(10):1281-8. doi: 10.1176/appi.ajp.2008.07121900. Epub 2008 Jun 16. PMID 18558642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from patients referred to the eating disorders program at The Ottawa Hospital by a family physician or psychiatrist between September 2000 and April 2006.
Groups:
- Placebo Plus Day Hospital: After a 2-week baseline period, placebo was administered for 10 weeks (weeks 3-12 of the study). Day hospital program involved attendance 4 days a week from 9:00 am to 6:00 pm for 12 to 14 weeks, and supervised meals and group therapy.
  Day Hospital: Day hospital program involved attendance 4 days a week from 9:00 am to 6:00 pm for 12 to 14 weeks, and supervised meals and group therapy.
Period: Overall Study
Arm/Group | Placebo Plus Day Hospital | Olanzapine Plus Day Hospital
Started | 18 | 16
Completed | 14 | 14
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Day Hospital | Olanzapine Plus Day Hospital | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.67 (11.59) | 23.61 (6.5) | 27.03 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI) (kg/m^2)
Description: Body Mass Index (BMI) measured in kg/m^2 units. Measured at Baseline (week 2) and post-treatment (week 13).
Time Frame: Baseline (week 2) and post-treatment (week 13)
Population: 4 participants discontinued in placebo group and 2 did not have weight measurements at week 13. 2 participants discontinued in the olanzapine group
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo Plus Day Hospital | Olanzapine Plus Day Hospital
Number analyzed (Participants) | 12 | 16
kg/m^2
  Week 2 baseline | 19.66 (1.32) | 20.30 (0.99)
  Week 13: number analyzed (Participants) | 12 | 14
  Week 13 | 19.66 (1.32) | 20.30 (0.99)

2. Secondary Outcome: Obsessions
Description: Obsessions subscale of the Yale-Brown Obsessive Compulsive Scale. Minimum score is 0 and maximum score is 20. Higher scores indicate higher levels of obsessions.
Time Frame: Pretreatment (Week 1) and Posttreatment (Week 13)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Plus Day Hospital | Olanzapine Plus Day Hospital
Number analyzed (Participants) | 18 | 16
units on a scale
  Pretreatment | 9.11 (5.58) | 11.06 (3.96)
  Posttreatment | 5.86 (4.83) | 6.54 (4.29)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Placebo Plus Day Hospital | Olanzapine Plus Day Hospital
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No